CLINICAL TRIAL: NCT01598571
Title: A Study to Assess the Absolute Bioavailability of a Single Oral Dose of Fostamatinib With Respect to an Intravenous Micro Tracer Dose of [14C] R406 in Healthy Male Volunteers
Brief Title: Study in Healthy Males to Assess Bioavailability of Single Fostamatinib With iv Micro Tracer Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00027; QBR112696
Record Dates: First submitted 2012-04-05; First posted 2012-05-15 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Healthy
Keywords: Phase 1; Healthy male volunteers; pharmacokinetics; fostamatinib; Bioavailability; R406 plasma AUC and Cmax; R406 plasma AUC0-t; t1/2λz; tmax
MeSH Terms: interventions — fostamatinib

ARMS (2):
- Fostamatinib 50 mg tablet (Experimental)
  Interventions: Drug: Fostamatinib
- Fostamatinib 100 μg [14C] R406 intravenous micro tracer dose (Experimental)
  Interventions: Drug: Fostamatinib

INTERVENTIONS:
Drug: Fostamatinib — Fostamatinib 50 mg tablet
  Arms: Fostamatinib 50 mg tablet
Drug: Fostamatinib — Fostamatinib 100 μg [14C] R406 intravenous micro tracer dose
  Arms: Fostamatinib 100 μg [14C] R406 intravenous micro tracer dose

SUMMARY:
Study in healthy males to assess bioavailability of single fostamatinib with iv micro tracer dose.

DETAILED DESCRIPTION:
A Study to Assess the Absolute Bioavailability of a Single Oral Dose of Fostamatinib with Respect to an Intravenous Micro Tracer Dose of [14C] R406 in Healthy Male Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18 to 55 years (inclusive), with a weight of at least 50 kg and a body mass index (BMI) between 18 and 30 kg/m2 (inclusive)
* Male volunteers willing to use barrier contraception ie, condoms with spermicide, from the first day of the investigational product administration until 3 months after the last administration of the investigational product

Exclusion Criteria:

* History of any clinically significant disease or disorder
* History or presence of GI, hepatic, or renal disease or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of drug
* Volunteers who smoke more than 5 cigarettes or the equivalent in tobacco per day
* Any clinically significant abnormalities in clinical chemistry, hematology or urinalysis results as judged by the Investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The percent of absolute bioavailability (F) of R406 after oral administration of fostamatinib. | Up to 96 hours post dose
Total radioactivity of [14C] R406 after an intravenous infusion of [14C]R406 in terms of AUC, AUC(0-t), Cmax, t1/2λz, MRT, CL, Vz. | Up to 96 hours post dose
  AUC-Area under the plasma concentration time curve; AUC(0-t)-Area under plasma concentration time curve from zero to time of the last measurable concentration; Cmax - max plasma concentration; t½ λz-Terminal half-life; MRT- Mean residence time; CL - Total body clearance; Vz - Volume of distribution during the terminal phase
Pharmacokinetic (PK) profile of a single oral dose of fostamatinib and a radiolabelled intravenous micro tracer dose of [14C] R406. | 0, 30min, 1h, 1h 30min, 1h 45min, 1h 50min, 1h 55min, 2, 2h 5min, 2h 10min, 2h 15min, 2h30min, 3, 3h 30min, 5h30min, 9h, 12h, 18h, 24h, 30h, 48h, 72h, 96h post-dose
  PK Parameters: AUC, AUC (0-t), Cmax, t½ λz and MRT

SECONDARY OUTCOMES:
Number of participants with Adverse Events. | Up to Day 12
Safety profile in terms of vital signs (blood pressure and pulse), clinical laboratory tests, ECGs and physical examination findings. | Up to Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Mark Layton, MD, Study Director — AstraZeneca, Alderley Park; Sharan Sidhu, MB CHB, BAO, MRCS, Principal Investigator — Quotient Clinical Unit
Locations (1):
- Ruddington, Nottingham, United Kingdom